CLINICAL TRIAL: NCT06352515
Title: Peripheral Blood T Lymphocyte Subsets in Ulcerative Colitis
Brief Title: T Lymphocyte Subsets in Ulcerative Colitis
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amany Abdelkader Ahmed, Assistant Lecturer, Assiut University
Other Study IDs: T cells in Ulcerative colitis
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Flow Cytometry

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serum sample will be stored at -70
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group I: Patients with newly diagnosed, active, untreated ulcerative colitis
  Interventions: Diagnostic Test: Flow cytometry
- Group II: Ulcerative colitis patients on non-biologic immunosuppressive drugs.
  Interventions: Diagnostic Test: Flow cytometry
- Group III: Ulcerative colitis patients on established biological treatment.
  Interventions: Diagnostic Test: Flow cytometry
- Group IV: Age- and sex-matched healthy controls.
  Interventions: Diagnostic Test: Flow cytometry

INTERVENTIONS:
Diagnostic Test: Flow cytometry — flow cytometry to study distribution of T lymphocyte subsets in ulcerative colitis patients

SUMMARY:
1. Study the distribution of peripheral blood T lymphocyte subsets among ulcerative colitis patients.
2. Correlation of T-cell subsets to therapeutic response/ disease activity.
3. Assess the value of circulating IgG anti-Integrin αvβ6 in UC.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is an idiopathic, chronic inflammatory disease of the large intestine, frequently involving the rectum, and characterized by chronic and recurrent mucosal inflammation and ulceration. Although its cause is not well understood, current evidence suggests innate and adaptive immunity play critical roles in its pathogenesis.

One of the main classes of immune cells that are affected by and contribute to UC is T cells. T-lymphocytes comprise a complex collection of highly differentiated T-cell subsets playing key roles in the regulation and the effector phase of the immune response. CD4+ T cells were found over-activated and proliferated in UC patients, which can induce disorders of the cytokine network and increase the occurrence of colitis.

Once intestinal pathogens or inflammatory mediators are not cleared in time, pro-inflammatory mononuclear phagocytes (MNPs) or polymorphonuclear leukocytes (PMNs) are often recruited to promote the polarization of naive CD4+ T cells into Th1, Th2, Th17, Treg and other subsets of cells.

The balances Th17/ Treg cells are important for maintaining intestinal homeostasis. Once the proportion Th17 cells increases, it often induces the production of pro-inflammatory cytokines that promote colonic inflammation, whereas Treg cells are usually secrete interleukin-10 (IL-10) and transforming growth factor-β (TGF-β) for anti-inflammatory regulations.

UC-associated inflammation is also characterized by huge number of activated B cells and plasma cells, the latter being involved in the production of cytotoxic granules, immunoglobulins, and various autoantibodies, Recent studies have highlighted a novel autoantibody against integrin αvβ6 in the serum of patients diagnosed with UC.

Recently, targeting immune cells to inhibit inflammation has become a research hotspot. Biological therapies are highly effective hallmark therapies in UC. Despite their widespread use, the impact of these agents on the composition of the adaptive immune system is largely unexplored. Knowledge on such effects in UC could clarify the mechanism of action of these therapies, provide information about the status of the adaptive immune system, and could help finding cell-based markers.

ELIGIBILITY:
Inclusion Criteria:

* patients with clinical diagnosis of ulcerative colitis among both sexes.
* Age >18 years Old.

Exclusion Criteria:

* Age <18 years old.
* Patients who refuse to participate in the study.
* Patients who have other autoimmune disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient >18 years diagnosed with ulcerative colitis including newly diagnosed patients, patients on non-biologic immunosuppressive drugs, and patients on biological treatment.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Study the distribution of T-cell subsets among ulcerative colitis patients. | 3 years
  Investigate and compare the distribution of different T-lymphocyte subsets among ulcerative colitis patients and healthy subjects .
Correlation of T-cell subtypes to therapeutic response | 3 years
  Determine the effect of different treatment strategies used in UC on T-lymphocyte subsets

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Abdelwahab, Study Director — Assiut University; Asmaa Bakr, Study Director — Assiut University; Tarek Elmelegy, Study Director — Assiut University

REFERENCES:
- [Background] Adolph TE, Meyer M, Schwarzler J, Mayr L, Grabherr F, Tilg H. The metabolic nature of inflammatory bowel diseases. Nat Rev Gastroenterol Hepatol. 2022 Dec;19(12):753-767. doi: 10.1038/s41575-022-00658-y. Epub 2022 Jul 29. PMID 35906289
- [Background] Huang J, Wang F, Tang X. Uncovering the shared molecule and mechanism between ulcerative colitis and atherosclerosis: an integrative genomic analysis. Front Immunol. 2023 Aug 10;14:1219457. doi: 10.3389/fimmu.2023.1219457. eCollection 2023. PMID 37638002
- [Background] Fan Q, Dai W, Li M, Wang T, Li X, Deng Z, Li W, Li M. Inhibition of alpha2,6-sialyltransferase relieves symptoms of ulcerative colitis by regulating Th17 cells polarization. Int Immunopharmacol. 2023 Dec;125(Pt A):111130. doi: 10.1016/j.intimp.2023.111130. Epub 2023 Oct 26. PMID 37897948
- [Background] Hua Y, Liu R, Lu M, Guan X, Zhuang S, Tian Y, Zhang Z, Cui L. Juglone regulates gut microbiota and Th17/Treg balance in DSS-induced ulcerative colitis. Int Immunopharmacol. 2021 Aug;97:107683. doi: 10.1016/j.intimp.2021.107683. Epub 2021 Apr 26. PMID 33915494
- [Background] Yang W, Liu H, Xu L, Yu T, Zhao X, Yao S, Zhao Q, Barnes S, Cohn SM, Dann SM, Zhang H, Zuo X, Li Y, Cong Y. GPR120 Inhibits Colitis Through Regulation of CD4+ T Cell Interleukin 10 Production. Gastroenterology. 2022 Jan;162(1):150-165. doi: 10.1053/j.gastro.2021.09.018. Epub 2021 Sep 16. PMID 34536451
- [Background] Saez A, Gomez-Bris R, Herrero-Fernandez B, Mingorance C, Rius C, Gonzalez-Granado JM. Innate Lymphoid Cells in Intestinal Homeostasis and Inflammatory Bowel Disease. Int J Mol Sci. 2021 Jul 16;22(14):7618. doi: 10.3390/ijms22147618. PMID 34299236
- [Background] Marafini I, Laudisi F, Salvatori S, Lavigna D, Venuto C, Giannarelli D, Monteleone G. Diagnostic value of anti-integrin alphavbeta6 antibodies in ulcerative colitis. Dig Liver Dis. 2024 Jan;56(1):55-60. doi: 10.1016/j.dld.2023.06.024. Epub 2023 Jul 6. PMID 37407314
- [Background] Dulic S, Toldi G, Sava F, Kovacs L, Molnar T, Milassin A, Farkas K, Rutka M, Balog A. Specific T-Cell Subsets Can Predict the Efficacy of Anti-TNF Treatment in Inflammatory Bowel Diseases. Arch Immunol Ther Exp (Warsz). 2020 Apr 4;68(2):12. doi: 10.1007/s00005-020-00575-5. PMID 32248339